CLINICAL TRIAL: NCT04151511
Title: "Continuous Thoracic Epidural Analgesia Versus Continuous Erector Spinae Plane Block for Postoperative Analgesia in Patients Undergoing Adult Living Donar Open Hepatectomies."
Brief Title: Continuous Thoracic Epidural Versus Erector Spinae Plane Block for Postoperative Analgesia in Donar Hepatectomies.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shifa Clinical Research Center (Other)
Collaborators: Shifa International Hospital (Other)
Responsible Party: Principal Investigator, Dr Muhammad Zubair, Associate Consultant Anaesthesiology, Shifa Clinical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB Ref #165-665-2019
Record Dates: First submitted 2019-10-22; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Thoracic Epidural (Other): Continuous Thoracic Epidural Analgesia for Postoperative Analgesia in Patients Undergoing Adult Living Donar Open Hepatectomies
  Interventions: Procedure: Continuous Erector Spinae Plane Block
- Continuous Erector Spinae Plane Block (Experimental): Continuous Erector Spinae Plane Block for Postoperative Analgesia in Patients Undergoing Adult Living Donar Open Hepatectomies
  Interventions: Procedure: Continuous Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Continuous Erector Spinae Plane Block — 1. Continuous Thoracic Epidural Thoracic Epidural Analgesia
  2. Continuous Erector Spinae Plane Block

SUMMARY:
Introduction Adult living related donor hepatectomy is associated with pain due to the sub-costal j-shaped incision, rib retraction using Thompson retractor, and diaphragm irritation1. The incidence of severe pain after donor hepatectomy is 11 to 37%2. Therefore adequate analgesia is important for optimum perioperative safety profiles and speedy recovery. Poor pain management is associated with risk of atelectasis, respiratory failure, and delayed discharge from the hospital.

so this study is comparison of two technique (Thoracic epidural analgesia vs Erector spinae plane block) to relieve pain.

DETAILED DESCRIPTION:
Thoracic epidural analgesia (TEA) is commonly used for pain management in donor hepatectomies. TEA reduces activation of the sympathetic outflow, surgical stress response, and pain-associated tachycardia and hypertension which can cause perioperative myocardial ischemia. TEA decreases stress-induced gastrointestinal disruption, immunosuppression, and decreases postoperative opioid requirement. TEA promotes expiratory intercostal and abdominal muscle tone and facilitates diaphragmatic excursion thus reduce the risks of atelectasis, pneumonia, and respiratory failure. However, TEA has its own drawbacks, e.g. hypotension caused by the inhibition of the sympathetic outflow, which can be associated with the administration of large amounts of crystalloids and colloids. Other complications may include failure to produce analgesia in 20% of patients3, intravascular cannulation leading to local anesthetic toxicity, unintentional dural punctures, paraesthesia, post-operative coagulopathies, epidural abscess, and epidural hematomas resulting in paraplegia1, 3. Considering these merits and demerits, TEA is the widely accepted choice for postoperative analgesia in living related donor hepatectomies1, 3,4, 5.

Erector spinae plane block (ESPB) is a novel ultrasound-guided regional anesthesia technique described in 2016 6 for the management of thoracic and abdominal pain. Ultrasound guidance is used to inject a local anesthetic in the interfacial plane between the erector spinae muscle and the associated transverse process of the spine. The mechanism of action is by the spread of local anesthetic anteriorly to the dorsal and ventral rami of the thoracic and abdominal spinal nerves 7. The absence of blood vessels in this vicinity shows the usefulness of this technique in the patients, who are prone to coagulopathies making it safer with lesser expertise, and with less procedural complications 8. The ESPB is an avascular plane block therefore, it results in lower plasma volumes rise due to reduced uptake of the local anesthetic by plasma hence the duration of action of local anesthetic is long. An ESPB at T5 level is sufficient to have a unilateral multi-dermatomes sensory block ranging from T1 to L3 level10 when used as a continuous block. Various case reports demonstrate its efficacy in a wide spectrum of specialities like acute and chronic pain management, thoraco-abdominal surgeries, neuropathic and post-traumatic pain 4, 7, 8,9 , 10. A comparison of continuous epidural versus single shot intrathecal morphine was made and assessed the quality of analgesia by a visual analog scale (VAS) and the additional IV analgesic requirements were 56% in cases of epidural 11 used for sample size calculation.

However, no randomized control study has been performed to compare the efficacy of a continuous ESPB with that of a continuous TEA for living related donor hepatectomies. Thus the aim of this study is to compare the postoperative analgesic efficacy and adverse effects of continuous ESPB to that of a continuous TEA in patients undergoing adult living donor hepatectomies. Investigators have hypothesized that continuous ESPB would provide better postoperative analgesia with fewer adverse effects. The primary outcome is post-operative pain scores using the visual analog scale (V.A.S) for pain at rest and at maximal inspiration during the post-operative period at PACU, 1, 6, 12, 24 and 48 hours. The secondary outcomes include lung incentive spirometry volumes, the dosage of adjunct nalbuphine used, hypotension, tachycardia, post-operative coagulopathy, early mobilization and discharge from surgical I.C.U (S.I.C.U).

Methodology After approval from the institutional and ethical review board and written informed consent, patients were randomized into either the TEA group or the ESPB group using the sealed enveloped method.

Study design The study will be a single-blinded, prospective, comparative, randomized control trial. The participants will be assigned to one of two groups; Group A will include patients receiving continuous TEA, whilst Group B will include patients receiving continuous ESPB. Both groups will receive their respective intervention after induction with standard general anesthesia.

Blinding is done at the level of assessor. The primary assessor will be blind with the type of technique applied and fill the Proforma according to standard routine with the same drug infusion.

Study population The study will include all adult patients undergoing elective living related donor hepatectomies for liver transplant surgery.

Study setting Study will be conducted in the liver transplant operating rooms of Shifa International Hospital.

Study duration The study duration will be of up to 12 months from the date of approval of the study from the hospital's institutional and ethical review board.

Randomization Randomization will be done by the simple random sampling technique using the sealed envelope method.

Sample Size Sample size was calculated by the WHO sample size calculator and using the following parameters; Level of significance - 5% Power of the test - 80% Proportion of patients requiring opioid in epidural group - 0.56 (ref no.13) Anticipated proportion of patients requiring opioid in ESP group - 0.25 Sample size - 30 patients in each group

Induction of General Anaesthesia In the operating room, the patient will be positioned on the operating table; the standard monitors: non-invasive blood pressure, ECG, pulse oximetry will be applied. A 20 gauge intravenous cannula will be secured on the dorsum of the hand and connected to a maintenance intravenous fluid therapy. The patient will be pre-oxygenated for 3 minutes with oxygen. The patient will be administered injection Ondansetron (0.1mg/kg) and injection Midazolam (0.02mg/kg) intravenous to start with. The patient will be induced with injection Buprenorphine (0.02mg/kg) and injection Propofol (2 mg/kg) mixed with Lidocaine (60 mg), and atracurium (0.5 mg/kg), after which an endotracheal tube will be inserted and mechanical ventilation will be initiated. A radial arterial line and a central venous line will be inserted. Both TEA and ESPB catheters will be placed after induction of general anesthesia for surgery by experienced practitioners in the left lateral decubitus position.

Data Collection Data for the study will be collected by a standardized performa which will record all the required variables of the study. Confidentiality of patient's data will be maintained.

Data Analysis The data will be analyzed by using the IBM SPSS software, version 25.0, for Windows.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 45 years of age
* A.S.A scores I - II Exclusion Criteria
* Neurological impairment
* Allergy, hypersensitivity or any other contraindications to local anesthetic
* Anatomical variation for block landmarks

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-19 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain scores | 6 hour
  Post-operative pain scores using the visual analog scale (V.A.S) 0-10 for pain at rest and at maximal inspiration during the post-operative period at PACU. 0 means no pain and 10 means unbearable pain. Higher scores would be worse outcome. primary outcome post-operative pain scores measured at 6 hours.

SECONDARY OUTCOMES:
The dosage of adjunct nalbuphine used (mg) | 6 hour
  The dosage of adjunct nalbuphine in milligrams (mg) required by the patient at 6 hours post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Muhammad Zubair, Principal Investigator — Shifa International Hospital
Locations (1):
- Hospital, Islamabad, Pakistan

REFERENCES:
- [Result] Kostov S, Schug SA. Depression and chronic pain. Saudi J Anaesth. 2018 Jul-Sep;12(3):377-378. doi: 10.4103/sja.SJA_69_18. No abstract available. PMID 30100833
- [Result] Dewe G, Steyaert A, De Kock M, Lois F, Reding R, Forget P. Pain management in living related adult donor hepatectomy: feasibility of an evidence-based protocol in 100 consecutive donors. BMC Res Notes. 2018 Nov 26;11(1):834. doi: 10.1186/s13104-018-3941-1. PMID 30477577
- [Result] Tzimas P, Prout J, Papadopoulos G, Mallett SV. Epidural anaesthesia and analgesia for liver resection. Anaesthesia. 2013 Jun;68(6):628-35. doi: 10.1111/anae.12191. PMID 23662750
- [Result] Chhibber A, Dziak J, Kolano J, Norton JR, Lustik S. Anesthesia care for adult live donor hepatectomy: our experiences with 100 cases. Liver Transpl. 2007 Apr;13(4):537-42. doi: 10.1002/lt.21074. PMID 17394151
- [Result] El-Boghdadly K, Pawa A. The erector spinae plane block: plane and simple. Anaesthesia. 2017 Apr;72(4):434-438. doi: 10.1111/anae.13830. Epub 2017 Feb 11. No abstract available. PMID 28188611
- [Result] Tsui BCH, Fonseca A, Munshey F, McFadyen G, Caruso TJ. The erector spinae plane (ESP) block: A pooled review of 242 cases. J Clin Anesth. 2019 Mar;53:29-34. doi: 10.1016/j.jclinane.2018.09.036. Epub 2018 Oct 3. PMID 30292068
- [Result] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Result] Jain K, Jaiswal V, Puri A. Erector spinae plane block: Relatively new block on horizon with a wide spectrum of application - A case series. Indian J Anaesth. 2018 Oct;62(10):809-813. doi: 10.4103/ija.IJA_263_18. PMID 30443066
- [Result] Adhikary SD, Pruett A, Forero M, Thiruvenkatarajan V. Erector spinae plane block as an alternative to epidural analgesia for post-operative analgesia following video-assisted thoracoscopic surgery: A case study and a literature review on the spread of local anaesthetic in the erector spinae plane. Indian J Anaesth. 2018 Jan;62(1):75-78. doi: 10.4103/ija.IJA_693_17. PMID 29416155
- [Result] Tulgar S, Selvi O, Kapakli MS. Erector Spinae Plane Block for Different Laparoscopic Abdominal Surgeries: Case Series. Case Rep Anesthesiol. 2018 Feb 18;2018:3947281. doi: 10.1155/2018/3947281. eCollection 2018. PMID 29670771
- [Result] De Pietri L, Siniscalchi A, Reggiani A, Masetti M, Begliomini B, Gazzi M, Gerunda GE, Pasetto A. The use of intrathecal morphine for postoperative pain relief after liver resection: a comparison with epidural analgesia. Anesth Analg. 2006 Apr;102(4):1157-63. doi: 10.1213/01.ane.0000198567.85040.ce. PMID 16551916
- [Derived] Zubair M, Adil Khan M, Khan MNA, Iqbal S, Ashraf M, Saleem SA. Comparison of Continuous Thoracic Epidural With Erector Spinae Block for Postoperative Analgesia in Adult Living Donor Hepatectomy. Cureus. 2022 Mar 14;14(3):e23151. doi: 10.7759/cureus.23151. eCollection 2022 Mar. PMID 35444875